CLINICAL TRIAL: NCT01038479
Title: Maternal Consumption of Xylitol to Reduce Early Childhood Decay (MaXED Study)
Acronym: MaXED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Fife (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Mr Brett Duane, NHS Fife
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09/S0501/49
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2009-12

CONDITIONS: Dental Caries; Oral Microbial Colonization
Keywords: Xylitol; Mutans streptococci; Maternal consumption; Early childhood tooth decay; Early childhood caries; Childsmile
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Childsmile programme with xylitol (Active Comparator): Childsmile program with maternal xylitol consumption;
  Interventions: Dietary Supplement: Xylitol consumption; Behavioral: Childsmile preventative programme
- Childsmile programme only (Placebo Comparator): Childsmile programme
  Interventions: Behavioral: Childsmile preventative programme

INTERVENTIONS:
Dietary Supplement: Xylitol consumption — Mothers will eat 6 grams of xylitol per day
  Arms: Childsmile programme with xylitol
Behavioral: Childsmile preventative programme — Mothers will receive the childsmile preventative programme
  Other Names: Mothers will receive the childsmile preventative programme

SUMMARY:
The purpose of this study is to determine if the Childsmile programme (www.child-smile.org) with the additional maternal use of xylitol is more effective at reducing dental decay in children than a Childsmile program alone.

The children will be compared in the two groups at age two, to determine how the interventions affected the early colonization of mutans streptococci, an important risk factor of tooth decay.

At three and at five years the investigators will also examine the amount of tooth decay in these children.

Using MIDAS (Scotland's national health service dental data) records, the investigators will follow the oral health of the children until the age of 5 years.

Main hypothesis:

The maternal consumption of xylitol reduces early childhood caries

DETAILED DESCRIPTION:
Xylitol has been shown to decrease mutans streptococci transmission between mother and child. Such maternal consumption of xylitol studies have, however not been tested in a Scottish population.

Sign 83, (www.sign.ac.uk/pdf/sign83.pdf) a Scottish government publication states that carrying out research in this area is needed.

Childsmile (www.child-smile.org) is a Scottish government programme that promotes oral health from birth, particularly amongst people living in priority areas.

Parents of newborn children who are assessed to be at risk of developing tooth decay are referred to the programme by their Health Visitor. Parents are visited at home by a Dental Health Support Worker. The dental health support worker will give more information, advice and arrange regular visits for participants to their local Dental Practice.

This research study will compare two groups; one group randomised into the childsmile preventative programme, the other group randomised into the childsmile preventative programme plus consuming 5 grams of xylitol per day.

We will be testing the mutans streptococci of the mother, at start of the study, and testing the mutans streptococci of mother and child at (child) aged two, in both groups- We will then be testing the dental decay of children in both groups

The research study will use existing NHS fife funding. NHS Fife currently employs approximately 15 dental health support workers, of which part of their role will be to support this project

Recruiting of study is planned to start in January 2010.

ELIGIBILITY:
Inclusion Criteria:

* Mother with high counts of MS (MS equal or higher than log 5)
* Child less than 3 months of age
* Has a close relationship with Fife (e.g. lives or works in Fife)
* Child seen by health visitor
* Mother who is the main carer of her children

Exclusion Criteria:

* Mother with low or no MS
* Child older than 3 months of age
* Child not seen by health visitor
* No close relationship with Fife (e.g. doesn't live or work in Fife)
* Mother who is not the main carer of her children

Ages: 2 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1064 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Caries occurrence at the age 3 and 5 yrs; | 5 years
Oral microbial colonization at 2 yrs | 2 years

SECONDARY OUTCOMES:
To determine the compliance and acceptability of xylitol consumption by the mother • Acceptability by the mother (as measured qualitatively using periodic questionnaires) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brett Duane, BDS,MAM, Principal Investigator — NHS Fife; Derek Richards, BDS MPH, Principal Investigator — NHS Forth Valley; Eva Soderling, PHD, Principal Investigator — University of Turku; Kaisu Pienihäkkinen, DDS, PhD, Principal Investigator — University of Turku
Locations (1):
- Brett Duane, NHS Fife, Leven, Fife, United Kingdom

REFERENCES:
- See also: Link to full protocol of study — http://www.nhsfife.scot.nhs.uk/CDS/approved%20full%20protocol%20V%206%5b1%5d.pdf